CLINICAL TRIAL: NCT03435081
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled, Phase 3 Study to Evaluate the Efficacy and Safety of Baricitinib in Adult Patients With Moderate to Severe Atopic Dermatitis
Brief Title: A Study of Baricitinib (LY3009104) in Adult Participants With Moderate to Severe Atopic Dermatitis
Acronym: BREEZE-AD5
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Collaborators: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 17049; I4V-MC-JAIW (Other: Eli Lilly and Company)
Record Dates: First submitted 2018-02-12; First posted 2018-02-15 (Actual); Results first posted 2021-01-25 (Actual); Last update posted 2022-09-09 (Actual); Status verified 2022-08

CONDITIONS: Atopic Dermatitis
Keywords: eczema; atopic eczema
MeSH Terms: conditions — Dermatitis, Atopic; Eczema | interventions — baricitinib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- 2 milligram (mg) Baricitinib (Experimental): 2 mg Baricitinib administered orally every day. Placebo administered orally to maintain the blind.
  Interventions: Drug: Baricitinib; Drug: Placebo
- 1 mg Baricitinib (Experimental): 1 mg Baricitinib administered orally every day. Placebo administered orally to maintain the blind.
  Interventions: Drug: Baricitinib; Drug: Placebo
- Placebo (Placebo Comparator): Placebo administered orally every day.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Baricitinib — Administered orally
  Other Names: LY3009104
  Arms: 1 mg Baricitinib; 2 milligram (mg) Baricitinib
Drug: Placebo — Administered orally

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of baricitinib in adult participants with moderate to severe atopic dermatitis.

ELIGIBILITY:
Inclusion Criteria:

* Have a diagnosis of atopic dermatitis (AD) at least 12 months before screening.
* Have moderate to severe AD, including all of the following:

  * EASI score ≥16
  * IGA score of ≥3
  * ≥10% of BSA involvement
* Have had inadequate response or intolerance to existing topical (applied to the skin) medications within 6 months preceding screening.
* Are willing to discontinue certain treatments for eczema (such as systemic and topical treatments during a washout period).
* Agree to use emollients daily.

Exclusion Criteria:

* Are currently experiencing or have a history of other concomitant skin conditions (e.g., psoriasis or lupus erythematosus), or a history of erythrodermic, refractory, or unstable skin disease that requires frequent hospitalizations and/or intravenous treatment for skin infections.
* A history of eczema herpeticum within 12 months, and/or a history of 2 or more episode of eczema herpeticum in the past.
* Participants who are currently experiencing a skin infection that requires treatment, or is currently being treated, with topical or systemic antibiotics.
* Have any serious illness that is anticipated to require the use of systemic corticosteroids or otherwise interfere with study participation or require active frequent monitoring (e.g., unstable chronic asthma).
* Have been treated with the following therapies:

  * monoclonal antibody for less than 5 half-lives before randomization
  * received prior treatment with any oral Janus kinase (JAK) inhibitor less than 4 weeks before randomization
  * received any parenteral corticosteroid administered by intramuscular or intravenous injection within 6 weeks of planned randomization or are anticipated to require parenteral injection of corticosteroids during the study
  * have had an intra-articular corticosteroid injection within 6 weeks of planned randomization
  * probenecid at the time of randomization that cannot be discontinued for the duration of the study
* Have high blood pressure characterized by a repeated systolic blood pressure >160 millimeters of mercury (mm Hg) or diastolic blood pressure >100 mm Hg.
* Have had major surgery within the past eight weeks or are planning major surgery during the study.
* Have experienced any of the following within 12 weeks of screening: myocardial infarction (MI), unstable ischemic heart disease, stroke, or New York Heart Association Stage III/IV heart failure.
* Have a history of venous thromboembolic event (VTE), or are considered at high risk for VTE.
* Have a history or presence of cardiovascular, respiratory, hepatic, chronic liver disease gastrointestinal, endocrine, hematological, neurological, lymphoproliferative disease or neuropsychiatric disorders or any other serious and/or unstable illness.
* Have a current or recent clinically serious viral, bacterial, fungal, or parasitic infection including herpes zoster, tuberculosis.
* Have specific laboratory abnormalities.
* Have received certain treatments that are contraindicated.
* Pregnant or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 440 (Actual)
Dates: Start 2018-02-20 (Actual); Primary Completion 2019-12-09 (Actual); Study Completion 2021-08-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (81):
- United States (60):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Johnson Dermatology, Fort Smith, Arkansas
  - Wallace Medical Group, Inc., Beverly Hills, California
  - California Dermatology and Clinical Research Institute, Encinitas, California
  - Tien Q. Nguyen, MD inc. DBA First OC Dermatology, Fountain Valley, California
  - Center for Dermatology Clinical Research, Inc., Fremont, California
  - Keck School of Medicine University of Southern California, Los Angeles, California
  - University of California Davis-Dermatology, Sacramento, California
  - Medical Center for Clinical Research, San Diego, California
  - University Clinical Trials, Inc., San Diego, California
  - Southern California Dermatology, Santa Ana, California
  - Clinical Science Institute, Santa Monica, California
  - Care Access Research-Walnut Creek, Walnut Creek, California
  - Clinical Research Center of CT/NY, Danbury, Connecticut
  - Univ of Connecticut, Farmington, Connecticut
  - GWU/Medical Faculty Associates, Washington D.C., District of Columbia
  - Solutions Through Advanced Research, Inc., Jacksonville, Florida
  - Olympian Clinical Research, Largo, Florida
  - Miami Dermatology & Laser Research, Miami, Florida
  - Riverchase Dermatology and Cosmetic Surgery, Pembroke Pines, Florida
  - University of South Florida, Tampa, Florida
  - ForCare Clinical Research, Tampa, Florida
  - Dermatologic Surgery Specialists, PC, Macon, Georgia
  - Advanced Medical Research, Sandy Springs, Georgia
  - Meridian Clinical Research, Savannah, Georgia
  - Treasure Valley Dermatology, Boise, Idaho
  - Northwestern University, Chicago, Illinois
  - University Dermatology, Darien, Illinois
  - Arlington Dermatology, Rolling Meadows, Illinois
  - Dawes Fretzin Clinical Research, Indianapolis, Indiana
  - The Indiana Clinical Trials Center, PC, Plainfield, Indiana
  - The South Bend Clinic, South Bend, Indiana
  - Dermatology Specialist, Louisville, Kentucky
  - Dermatology and Skin Cancer Specialists, Rockville, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - Brigham and Womens Hospital, Boston, Massachusetts
  - Great Lakes Research Group, Inc., Bay City, Michigan
  - Hamzavi Dermatology, Fort Gratiot, Michigan
  - Central Dermatology PC, St Louis, Missouri
  - Skin Specialists, P.C, Omaha, Nebraska
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - DermResearchCenter of New York, Inc, Stony Brook, New York
  - Bexley Dermatology Research, Bexley, Ohio
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Wright State Univ School of Medicine, Fairborn, Ohio
  - Dermatologists of Southwest Ohio, Inc., Mason, Ohio
  - Oregon Dermatology and Research Center, Portland, Oregon
  - OHSU Center for Health and Healing, Portland, Oregon
  - Dermatology and Skin Surgery Center, Exton, Pennsylvania
  - Clinical Partners LLC, Johnston, Rhode Island
  - Dermatology & Laser Center of Charleston, Charleston, South Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - Bellaire Dermatology, Bellaire, Texas
  - Modern Research Associates PLLC, Dallas, Texas
  - Austin Institute for Clinical Research, Inc., Pflugerville, Texas
  - Texas Dermatology and Laser Specialists, San Antonio, Texas
  - Acclaim Dermatology, PLLC, Sugar Land, Texas
  - University of Utah MidValley Dematology, Murray, Utah
  - Virginia Clinical Research, Norfolk, Virginia
  - Multicare Health System, Tacoma, Washington
- Canada (17):
  - Kirk Barber Research, Calgary, Alberta
  - Institute for Skin Advancement, Calgary, Alberta
  - Stratica Medical, Edmonton, Alberta
  - Dr. Chih-ho Hong Medical Inc., Surrey, British Columbia
  - Enverus Medical Research, Surrey, British Columbia
  - Simcoderm Medical & Surgical Dermatology Centre, Barrie, Ontario
  - Kingsway Clinical Research, Etobicoke, Ontario
  - Medicor Research Inc, Greater Sudbury, Ontario
  - Lynderm Research Inc, Markham, Ontario
  - Allergy Research Canada Inc., Niagara Falls, Ontario
  - SKiN Centre for Dermatology, Peterborough, Ontario
  - The Centre for Dermatology, Richmond Hill, Ontario
  - K. Papp Clinical Research Inc, Waterloo, Ontario
  - XLR8 Medical Research, Windsor, Ontario
  - Innovaderm Research Inc, Montreal, Quebec
  - Centre de Recherche Dermatologique de Quebec Metropolitain, Québec, Quebec
  - York Dermatology Center, Richmond Hill
- Puerto Rico (4):
  - Office of Dr. Samuel Sanchez PSC, Caguas, PR
  - Office of Dr. Alma M. Cruz, Carolina, PR
  - Ponce School of Medicine CAIMED Center, Ponce, PR
  - GCM Medical Group PSC, San Juan, PR

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

REFERENCES:
- [Derived] Wollenberg A, Kircik L, Simpson E, Brinker D, Katoh N, Rueda MJ, Issa M, Yang F, Feely M, Alexis A. Pooled Analysis of Baricitinib Tolerability in Patients With Atopic Dermatitis in Relation to Acne, Headache, and Gastrointestinal Events From 8 Clinical Trials. Dermatitis. 2023 Jul-Aug;34(4):308-314. doi: 10.1089/derm.2022.0027. Epub 2023 Feb 6. PMID 36749121
- [Derived] Simpson EL, Bissonnette R, Paller AS, King B, Silverberg JI, Reich K, Thyssen JP, Doll H, Sun L, DeLozier AM, Nunes FP, Eichenfield LF. The Validated Investigator Global Assessment for Atopic Dermatitis (vIGA-AD): a clinical outcome measure for the severity of atopic dermatitis. Br J Dermatol. 2022 Oct;187(4):531-538. doi: 10.1111/bjd.21615. Epub 2022 Aug 21. PMID 35442530
- [Derived] Rosmarin D, Casillas M, Chen S, Dawson Z, Pierce E, Zhang H, Bukhalo M, Smith S. Onset of Symptom Relief Reported in Daily Diaries of Patients With Atopic Dermatitis Treated With Baricitinib in a United States Clinical Trial (BREEZE-AD5). J Cutan Med Surg. 2022 May-Jun;26(3):262-266. doi: 10.1177/12034754211073661. Epub 2022 Jan 28. PMID 35086348
- [Derived] Silverberg JI, Boguniewicz M, Waibel J, Weisman J, Strowd L, Sun L, Ding Y, Feely M, Nunes FP, Simpson EL. Clinical Tailoring of Baricitinib 2 mg in Atopic Dermatitis: Baseline Body Surface Area and Rapid Onset of Action Identifies Response at Week 16. Dermatol Ther (Heidelb). 2022 Jan;12(1):137-148. doi: 10.1007/s13555-021-00640-7. Epub 2021 Nov 30. PMID 34846636
- [Derived] Silverberg JI, DeLozier A, Sun L, Thyssen JP, Kim B, Yosipovitch G, Nunes FP, Gugiu PC, Doll HA, Eichenfield LF. Psychometric properties of the itch numeric rating scale, skin pain numeric rating scale, and atopic dermatitis sleep scale in adult patients with moderate-to-severe atopic dermatitis. Health Qual Life Outcomes. 2021 Oct 23;19(1):247. doi: 10.1186/s12955-021-01877-8. PMID 34688290
- [Derived] King B, Maari C, Lain E, Silverberg JI, Issa M, Holzwarth K, Brinker D, Cardillo T, Nunes FP, Simpson EL. Extended Safety Analysis of Baricitinib 2 mg in Adult Patients with Atopic Dermatitis: An Integrated Analysis from Eight Randomized Clinical Trials. Am J Clin Dermatol. 2021 May;22(3):395-405. doi: 10.1007/s40257-021-00602-x. Epub 2021 Apr 7. PMID 33826132
- See also: A Study of Baricitinib (LY3009104) in Adult Participants With Moderate to Severe Atopic Dermatitis (Eczema) (BREEZE-AD5) — https://trials.lillytrialguide.com/en-US/trial/1Wc7bHopCgKYI4SqseaaSI

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants who did not meet IGA 0 or 1 at Week 16 and completed at least 16 Weeks in JAIW were discontinued and if eligible had the option to roll over into the Open-Label Extension study JAIX (NCT03559720).
Groups:
- 1 Milligram (mg) Baricitinib: 1 mg Baricitinib administered orally every day. Placebo administered orally to maintain the blind.
- 2 mg Baricitinib: 2 mg Baricitinib administered orally every day. Placebo administered orally to maintain the blind.
Period: Week 0 to Week 16
Arm/Group | Placebo | 1 Milligram (mg) Baricitinib | 2 mg Baricitinib
Started | 147 | 147 | 146
Received at Least One Dose of Study Drug | 147 | 147 | 146
Completed Week 16 and Entered JAIX Study | 111 | 112 | 96
Completed | 126 | 131 | 127
Not Completed | 21 | 16 | 19
Not completed — Lack of Efficacy | 6 | 5 | 0
Not completed — Adverse Event | 2 | 2 | 2
Not completed — Withdrawal by Subject | 8 | 7 | 10
Not completed — Lost to Follow-up | 3 | 1 | 4
Not completed — Pregnancy | 1 | 0 | 0
Not completed — Non-compliance | 1 | 0 | 2
Not completed — Inadequate Response | 0 | 1 | 0
Not completed — Withdrawal Due to Caregiver Circumstance | 0 | 0 | 1
Period: Week 16 to Week 104
Arm/Group | Placebo | 1 Milligram (mg) Baricitinib | 2 mg Baricitinib
Started | 8 (Participants who met IGA 0 or 1 and did not require rescue therapy before Week 16 were allowed to continue in the study beyond 16 weeks.) | 19 (Participants who met IGA 0 or 1 and did not require rescue therapy before Week 16 were allowed to continue in the study beyond 16 weeks.) | 35 (Participants who met IGA 0 or 1 and did not require rescue therapy before Week 16 were allowed to continue in the study beyond 16 weeks.)
Rolled Over Into the Open-Label Extension Study JAIX. | 6 (Participants who completed Week 104 and participants who experienced a loss of benefit (IGA score of ≥3) after Week 16, if eligible, had the option to roll over into the Open-Label Extension study JAIX.) | 14 (Participants who completed Week 104 and participants who experienced a loss of benefit (IGA score of ≥3) after Week 16, if eligible, had the option to roll over into the Open-Label Extension study JAIX.) | 19 (Participants who completed Week 104 and participants who experienced a loss of benefit (IGA score of ≥3) after Week 16, if eligible, had the option to roll over into the Open-Label Extension study JAIX.)
Completed | 5 | 6 | 16
Not Completed | 3 | 13 | 19
Not completed — Lack of Efficacy | 2 | 11 | 10
Not completed — Adverse Event | 1 | 0 | 2
Not completed — Withdrawal by Subject | 0 | 1 | 2
Not completed — Lost to Follow-up | 0 | 1 | 4
Not completed — Non--Compliance | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: All randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | 1 mg Baricitinib | 2 mg Baricitinib | Total
Number analyzed (Participants) | 147 | 147 | 146 | 440
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 134 | 134 | 137 | 405
  >=65 years | 13 | 13 | 9 | 35
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 67 | 72 | 77 | 216
  Male | 80 | 75 | 69 | 224
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 2 | 2 | 6
  Asian | 33 | 26 | 22 | 81
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 2 | 2
  Black or African American | 24 | 26 | 30 | 80
  White | 80 | 86 | 85 | 251
  More than one race | 7 | 6 | 5 | 18
  Unknown or Not Reported | 1 | 1 | 0 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 42 | 40 | 37 | 119
  United States | 105 | 107 | 109 | 321

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving Eczema Area and Severity Index 75 (EASI75) (2 mg Baricitinib)
Description: The EASI assesses objective physician estimates of 2 dimensions of atopic dermatitis - disease extent and clinical signs affected: 0 = 0%; 1 = 1-9%; 2 = 10-29%; 3 = 30-49%; 4 = 50-69%; 5 = 70-89%; 6 = 90-100% and the severity of 4 clinical signs: (1) erythema, (2) edema/papulation, (3) excoriation, and (4) lichenification each on a scale of 0 to 3 (0 = none, absent; 1 = mild; 2 = moderate; 3 = severe) at 4 body sites (head/neck, trunk, upper limbs, and lower limbs). Half scores are allowed between severities 1, 2, and 3. The final EASI score was obtained by weight-averaging these 4 scores and will range from 0 to 72 (severe). The EASI75 is defined as a ≥ 75% improvement from baseline in the EASI score.
Time Frame: Week 16
Population: All participants randomized to placebo or 2 mg of study drug. As pre-specified in the analysis plan, outcome measures will not be reported for the Maximum Extended Enrollment (MEE) arms/groups but only for the main global study arms/groups.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | 2 mg Baricitinib
Number analyzed (Participants) | 147 | 146
percentage of participants | 8.2 [4.7 to 13.7] | 29.5 [22.7 to 37.3]
Statistical Analysis 1: Comparison: Placebo vs 2 mg Baricitinib; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 4.60, 95% CI 2-sided [2.31 to 9.15]

2. Secondary Outcome: Percentage of Participants Achieving Investigator's Global Assessment (IGA) of 0 or 1 With a ≥ 2 Point Improvement
Description: The IGA measures the investigator's global assessment of the participant's overall severity of their AD, based on a static, numeric 5-point scale from 0 (clear skin) to 4 (severe disease). The score is based on an overall assessment of the degree of erythema, papulation/induration, oozing/crusting, and lichenification.
Time Frame: Week 16
Population: All randomized participants. As pre-specified in the analysis plan, outcome measures will not be reported for the Maximum Extended Enrollment (MEE) arms/groups but only for the main global study arms/groups.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | 1 mg Baricitinib | 2 mg Baricitinib
Number analyzed (Participants) | 147 | 147 | 146
percentage of participants | 5.4 [2.8 to 10.4] | 12.9 [8.4 to 19.3] | 24.0 [17.8 to 31.5]
Statistical Analysis 1: Comparison: Placebo vs 1 mg Baricitinib; Test type: Superiority; p = 0.033, Regression, Logistic; Odds Ratio (OR) = 2.51, 95% CI 2-sided [1.08 to 5.83]
Statistical Analysis 2: Comparison: Placebo vs 2 mg Baricitinib; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 5.29, 95% CI 2-sided [2.40 to 11.68]

3. Secondary Outcome: Percentage of Participants Achieving EASI75 (1 mg Baricitinib)
Description: as for outcome 1
Time Frame: Week 16
Population: All participants randomized to placebo or 1 mg of study drug. As pre-specified in the analysis plan, outcome measures will not be reported for the Maximum Extended Enrollment (MEE) arms/groups but only for the main global study arms/groups.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | 1 mg Baricitinib
Number analyzed (Participants) | 147 | 147
percentage of participants | 8.2 [4.7 to 13.7] | 12.9 [8.4 to 19.3]
Statistical Analysis 1: Comparison: Placebo vs 1 mg Baricitinib; Test type: Superiority; p = 0.167, Regression, Logistic; Odds Ratio (OR) = 1.71, 95% CI 2-sided [0.80 to 3.63]

4. Secondary Outcome: Percentage of Participants Achieving EASI90
Description: The EASI assesses objective physician estimates of 2 dimensions of atopic dermatitis - disease extent and clinical signs affected: 0 = 0%; 1 = 1-9%; 2 = 10-29%; 3 = 30-49%; 4 = 50-69%; 5 = 70-89%; 6 = 90-100% and the severity of 4 clinical signs: (1) erythema, (2) edema/papulation, (3) excoriation, and (4) lichenification each on a scale of 0 to 3 (0 = none, absent; 1 = mild; 2 = moderate; 3 = severe) at 4 body sites (head/neck, trunk, upper limbs, and lower limbs). Half scores are allowed between severities 1, 2, and 3. The final EASI score was obtained by weight-averaging these 4 scores and will range from 0 to 72 (severe). The EASI90 is defined as a ≥ 90% improvement from baseline in the EASI score.
Time Frame: Week 16
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | 1 mg Baricitinib | 2 mg Baricitinib
Number analyzed (Participants) | 147 | 147 | 146
percentage of participants | 3.4 [1.5 to 7.7] | 7.5 [4.2 to 12.9] | 20.5 [14.8 to 27.8]
Statistical Analysis 1: Comparison: Placebo vs 1 mg Baricitinib; Test type: Superiority; p = 0.131, Regression, Logistic; Odds Ratio (OR) = 2.23, 95% CI 2-sided [0.79 to 6.31]
Statistical Analysis 2: Comparison: Placebo vs 2 mg Baricitinib; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 6.73, 95% CI 2-sided [2.63 to 17.19]

5. Secondary Outcome: Percent Change From Baseline in EASI Score
Description: The EASI assesses objective physician estimates of 2 dimensions of atopic dermatitis - disease extent and clinical signs affected: 0 = 0%; 1 = 1-9%; 2 = 10-29%; 3 = 30-49%; 4 = 50-69%; 5 = 70-89%; 6 = 90-100% and the severity of 4 clinical signs: (1) erythema, (2) edema/papulation, (3) excoriation, and (4) lichenification each on a scale of 0 to 3 (0 = none, absent; 1 = mild; 2 = moderate; 3 = severe) at 4 body sites (head/neck, trunk, upper limbs, and lower limbs). Half scores are allowed between severities 1, 2, and 3. The final EASI score was obtained by weight-averaging these 4 scores and will range from 0 to 72 (severe).
  Least Squares (LS) Means were calculated using a MMRM model with treatment, baseline disease severity (IGA), visit, and treatment-by-visit-interaction as fixed categorical effects and baseline and baseline-by-visit-interaction as fixed continuous effects.
Time Frame: Baseline, Week 16
Population: All randomized participants with Week 16 EASI data. As pre-specified in the analysis plan, outcome measures will not be reported for the Maximum Extended Enrollment (MEE) arms/groups but only for the main global study arms/groups.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo | 1 mg Baricitinib | 2 mg Baricitinib
Number analyzed (Participants) | 28 | 47 | 62
percent change | -34.07 (5.529) | -46.66 (4.469) | -54.37 (4.156)
Statistical Analysis 1: Comparison: Placebo vs 1 mg Baricitinib; Test type: Superiority; p = 0.077, Mixed Models Analysis; Mean Difference (Final Values) = -12.59, 95% CI 2-sided [-26.54 to 1.36], Standard Error of Mean 7.079
Statistical Analysis 2: Comparison: Placebo vs 2 mg Baricitinib; Test type: Superiority; p = 0.004, Mixed Models Analysis; Mean Difference (Final Values) = -20.30, 95% CI 2-sided [-33.85 to -6.75], Standard Error of Mean 6.875

6. Secondary Outcome: Percentage of Participants Achieving SCORing Atopic Dermatitis 75 (SCORAD75)
Description: The SCORAD index uses the rule of nines to assess disease extent and evaluates 6 clinical characteristics to determine disease severity: (1) erythema, (2) edema/papulation, (3)oozing/crusts, (4) excoriation, (5) lichenification, and (6) dryness on a scale of 0 to 3 (0=absence, 1=mild, 2=moderate, 3=severe). The SCORAD index also assesses subjective symptoms of pruritus and sleep loss with a visual analogue scales (VAS) where 0 is no itching or no trouble sleeping and 10 is unbearable itching or a lot of trouble sleeping. These 3 aspects: extent of disease (A: 0-1-2), disease severity (B: 0-18), & subjective symptoms (C: 0-20) combine using A/5 + 7*B/2+ C to give a maximum possible score of 103, where 0 = no disease and 103 = severe disease. The SCORAD75 responder is defined as a participant who achieves a ≥ 75% improvement from baseline in the SCORAD score.
Time Frame: Week 16
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | 1 mg Baricitinib | 2 mg Baricitinib
Number analyzed (Participants) | 147 | 147 | 146
percentage of participants | 2.7 [1.1 to 6.8] | 3.4 [1.5 to 7.7] | 14.4 [9.6 to 21.0]
Statistical Analysis 1: Comparison: Placebo vs 1 mg Baricitinib; Test type: Superiority; p = 0.733, Regression, Logistic; Odds Ratio (OR) = 1.24, 95% CI 2-sided [0.36 to 4.36]
Statistical Analysis 2: Comparison: Placebo vs 2 mg Baricitinib; Test type: Superiority; p = 0.002, Regression, Logistic; Odds Ratio (OR) = 5.42, 95% CI 2-sided [1.93 to 15.22]

7. Secondary Outcome: Percentage of Participants Achieving a 4-Point Improvement on the Itch Numeric Rating Scale (NRS)
Description: The Itch NRS is a patient-administered, 11-point horizontal scale anchored at 0 and 10, with 0 representing "no itch" and 10 representing "worst itch imaginable." Overall severity of a participant's itching is indicated by selecting the number, using a daily diary, that best describes the worst level of itching in the past 24 hours.
Time Frame: 16 Weeks
Population: All randomized participants with a Baseline Itch NRS score >=4.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | 1 mg Baricitinib | 2 mg Baricitinib
Number analyzed (Participants) | 123 | 132 | 131
percentage of participants | 5.7 [2.8 to 11.3] | 15.9 [10.6 to 23.1] | 25.2 [18.5 to 33.3]
Statistical Analysis 1: Comparison: Placebo vs 1 mg Baricitinib; Test type: Superiority; p = 0.012, Regression, Logistic; Odds Ratio (OR) = 3.08, 95% CI 2-sided [1.29 to 7.36]
Statistical Analysis 2: Comparison: Placebo vs 2 mg Baricitinib; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 5.32, 95% CI 2-sided [2.31 to 12.28]

8. Secondary Outcome: Change From Baseline in the Score of Item 2 of the Atopic Dermatitis Sleep Scale (ADSS)
Description: Atopic Dermatitis Sleep Scale (ADSS) is a 3-item, participant-administered questionnaire developed to assess the impact of itch on sleep including difficulty falling asleep, frequency of waking, and difficulty getting back to sleep last night. Item 2, frequency of waking last night is reported by selecting the number of times they woke up each night, ranging from 0 to 29 times, where the higher a number indicates a worse outcome. The ADSS is designed to be completed daily, using a daily diary, with respondents thinking about sleep "last night." Each item is scored individually.
  LS Means were calculated using a MMRM model with treatment, region, baseline disease severity (IGA), visit, and treatment-by-visit-interaction as fixed categorical effects and baseline and baseline-by- visit-interaction as fixed continuous effects.
Time Frame: Baseline, Week 16
Population: All randomized participants with Week 16 ADSS Item 2 (frequency of waking) data.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | 1 mg Baricitinib | 2 mg Baricitinib
Number analyzed (Participants) | 37 | 64 | 73
units on a scale | -0.40 (0.207) | -0.62 (0.177) | -0.99 (0.171)
Statistical Analysis 1: Comparison: Placebo vs 1 mg Baricitinib; Test type: Superiority; p = 0.433, Mixed Models Analysis; Mean Difference (Final Values) = -0.21, 95% CI 2-sided [-0.75 to 0.32], Standard Error of Mean 0.273
Statistical Analysis 2: Comparison: Placebo vs 2 mg Baricitinib; Test type: Superiority; p = 0.029, Mixed Models Analysis; Mean Difference (Final Values) = -0.59, 95% CI 2-sided [-1.12 to -0.06], Standard Error of Mean 0.269

9. Secondary Outcome: Change From Baseline in Skin Pain NRS
Description: Skin Pain NRS is a participant-administered, 11-point horizontal scale anchored at 0 and 10, with 0 representing "no pain" and 10 representing "worst pain imaginable." Overall severity of a participant's skin pain is indicated by selecting the number, using a daily diary, that best describes the worst level of skin pain in the past 24 hours.
  LS Means were calculated using a MMRM model with treatment, baseline disease severity (IGA), visit, and treatment-by-visit-interaction as fixed categorical effects and baseline and baseline-by-visit-interaction as fixed continuous effects.
Time Frame: Baseline, Week 16
Population: All randomized participants with Week 16 Skin Pain NRS data.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | 1 mg Baricitinib | 2 mg Baricitinib
Number analyzed (Participants) | 37 | 64 | 73
units on a scale | -1.03 (0.342) | -2.16 (0.279) | -2.40 (0.266)
Statistical Analysis 1: Comparison: Placebo vs 1 mg Baricitinib; Test type: Superiority; p = 0.012, Mixed Models Analysis; Mean Difference (Final Values) = -1.12, 95% CI 2-sided [-1.99 to -0.25], Standard Error of Mean 0.441
Statistical Analysis 2: Comparison: Placebo vs 2 mg Baricitinib; Test type: Superiority; p = 0.002, Mixed Models Analysis; Mean Difference (Final Values) = -1.36, 95% CI 2-sided [-2.22 to -0.51], Standard Error of Mean 0.433

10. Secondary Outcome: Percentage of of Participants Achieving EASI50
Description: The EASI assesses objective physician estimates of 2 dimensions of atopic dermatitis - disease extent and clinical signs affected: 0 = 0%; 1 = 1-9%; 2 = 10-29%; 3 = 30-49%; 4 = 50-69%; 5 = 70-89%; 6 = 90-100%) and the severity of 4 clinical signs (erythema, edema/papulation, excoriation, and lichenification) each on a scale of 0 to 3 (0 = none, absent; 1 = mild; 2 = moderate; 3 = severe) at 4 body sites (head and neck, trunk, upper limbs, and lower limbs). Half scores are allowed between severities 1, 2 and 3. The final EASI score was obtained by weight-averaging these 4 scores and will range from 0 to 72 (severe). The EASI50 is defined as a ≥ 50% improvement from baseline in EASI score.
Time Frame: Week 16
Population: All randomized participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | 1 mg Baricitinib | 2 mg Baricitinib
Number analyzed (Participants) | 147 | 147 | 146
percentage of participants | 12.9 [8.4 to 19.3] | 19.7 [14.1 to 26.9] | 34.9 [27.7 to 43.0]
Statistical Analysis 1: Comparison: Placebo vs 1 mg Baricitinib; Test type: Superiority; p = 0.105, Regression, Logistic; Odds Ratio (OR) = 1.69, 95% CI 2-sided [0.90 to 3.20]
Statistical Analysis 2: Comparison: Placebo vs 2 mg Baricitinib; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 3.67, 95% CI 2-sided [2.02 to 6.68]

11. Secondary Outcome: Percentage of Participants Achieving IGA of 0
Description: as for outcome 2
Time Frame: Week 16
Population: All randomized participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | 1 mg Baricitinib | 2 mg Baricitinib
Number analyzed (Participants) | 147 | 147 | 146
percentage of participants | 0.7 [0.1 to 3.8] | 3.4 [1.5 to 7.7] | 2.7 [1.1 to 6.8]
Statistical Analysis 1: Comparison: Placebo vs 1 mg Baricitinib; Test type: Superiority; p = 0.144, Regression, Logistic; Odds Ratio (OR) = 3.81, 95% CI 2-sided [0.63 to 22.85]
Statistical Analysis 2: Comparison: Placebo vs 2 mg Baricitinib; Test type: Superiority; p = 0.227, Regression, Logistic; Odds Ratio (OR) = 3.10, 95% CI 2-sided [0.50 to 19.40]

12. Secondary Outcome: Change From Baseline in SCORAD
Description: The SCORAD index uses the rule of nines to assess disease extent and evaluates 6 clinical characteristics to determine disease severity: (1) erythema, (2) edema/papulation, (3) oozing/crusts, (4) excoriation, (5) lichenification, and (6) dryness on a scale of 0 to 3 (0=absence, 1=mild, 2=moderate, 3=severe). The SCORAD index also assesses subjective symptoms of pruritus and sleep loss with VAS where 0 is no itching or no trouble sleeping and 10 is unbearable itching or a lot of trouble sleeping. These 3 aspects: extent of disease (A: 0-1-2), disease severity (B: 0-18), & subjective symptoms (C: 0-20) combine using A/5 + 7*B/2+ C to give a maximum possible score of 103, where 0 = no disease and 103 = severe disease.
  LS Means were calculated using a MMRM model with treatment, baseline disease severity (IGA), visit and treatment-by-visit interaction as fixed categorial effects and baseline and baseline-by-visit interaction as fixed continuous effects.
Time Frame: Baseline, Week 16
Population: All randomized participants with Week 16 SCORAD data.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | 1 mg Baricitinib | 2 mg Baricitinib
Number analyzed (Participants) | 28 | 46 | 61
units on a scale | -14.37 (3.058) | -18.31 (2.445) | -26.18 (2.220)
Statistical Analysis 1: Comparison: Placebo vs 1 mg Baricitinib; Test type: Superiority; p = 0.316, Mixed Models Analysis; Mean Difference (Final Values) = -3.94, 95% CI 2-sided [-11.67 to 3.79], Standard Error of Mean 3.921
Statistical Analysis 2: Comparison: Placebo vs 2 mg Baricitinib; Test type: Superiority; p = 0.002, Mixed Models Analysis; Mean Difference (Final Values) = -11.81, 95% CI 2-sided [-19.23 to -4.40], Standard Error of Mean 3.758

13. Secondary Outcome: Percentage of Participants Achieving SCORAD90
Description: The SCORAD index uses the rule of nines to assess disease extent and evaluates 6 clinical characteristics to determine disease severity: (1) erythema, (2) edema/papulation, (3) oozing/crusts, (4) excoriation, (5) lichenification, and (6) dryness on a scale of 0 to 3 (0=absence, 1=mild, 2=moderate, 3=severe). The SCORAD index also assesses subjective symptoms of pruritus and sleep loss with VAS where 0 is no itching or no trouble sleeping and 10 is unbearable itching or a lot of trouble sleeping. These 3 aspects: extent of disease (A: 0-1-2), disease severity (B: 0-18), & subjective symptoms (C: 0-20) combine using A/5 + 7*B/2+ C to give a maximum possible score of 103, where 0 = no disease and 103 = severe disease. SCORAD90 is defined as a ≥ 90% improvement from baseline in the SCORAD score.
Time Frame: Week 16
Population: All randomized participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | 1 mg Baricitinib | 2 mg Baricitinib
Number analyzed (Participants) | 147 | 147 | 146
percentage of participants | 1.4 [0.4 to 4.8] | 2.0 [0.7 to 5.8] | 3.4 [1.5 to 7.8]
Statistical Analysis 1: Comparison: Placebo vs 1 mg Baricitinib; Test type: Superiority; p = 0.683, Regression, Logistic; Odds Ratio (OR) = 1.39, 95% CI 2-sided [0.29 to 6.78]
Statistical Analysis 2: Comparison: Placebo vs 2 mg Baricitinib; Test type: Superiority; p = 0.277, Regression, Logistic; Odds Ratio (OR) = 2.25, 95% CI 2-sided [0.52 to 9.68]

14. Secondary Outcome: Change From Baseline in Body Surface Area (BSA) Affected
Description: Body surface area affected by AD will be assessed for 4 separate body regions and is collected as part of the EASI assessment: head and neck, trunk (including genital region), upper extremities, and lower extremities (including the buttocks). Each body region will be assessed for disease extent ranging from 0% to 100% involvement. The overall total percentage will be reported based off of all 4 body regions combined, after applying specific multipliers to the different body regions to account for the percent of the total BSA represented by each of the 4 regions. Use the percentage of skin affected for each region (0 to 100%) in EASI as follows: BSA Total = 0.1*BSAhead and neck + 0.3*BSAtrunk + 0.2* BSAupper limbs + 0.4*BSAlower limbs.
  LS Means were calculated using a MMRM model with treatment, baseline disease severity (IGA), visit, and treatment-by-visit-interaction as fixed categorical effects and baseline and baseline-by-visit-interactions as fixed continuous effects.
Time Frame: Baseline, Week 16
Population: All randomized participants with Week 16 BSA data.
Measure: Least Squares Mean (Standard Error); unit: percentage of BSA
Arm/Group | Placebo | 1 mg Baricitinib | 2 mg Baricitinib
Number analyzed (Participants) | 28 | 47 | 62
percentage of BSA | -9.67 (2.352) | -15.69 (1.885) | -17.39 (1.746)
Statistical Analysis 1: Comparison: Placebo vs 1 mg Baricitinib; Test type: Superiority; p = 0.046, Mixed Models Analysis; Mean Difference (Final Values) = -6.02, 95% CI 2-sided [-11.93 to -0.12], Standard Error of Mean 2.996
Statistical Analysis 2: Comparison: Placebo vs 2 mg Baricitinib; Test type: Superiority; p = 0.009, Mixed Models Analysis; Mean Difference (Final Values) = -7.72, 95% CI 2-sided [-13.46 to -1.98], Standard Error of Mean 2.911

15. Secondary Outcome: Percentage of Participants Developing Skin Infections Requiring Antibiotic Treatment
Description: Percentage of participants developing skin infections requiring antibiotic treatment.
Time Frame: Week 16
Population: All randomized participants who received at least 1 dose of study drug and who did not discontinue from study for reason lost to follow-up at the first post-baseline visit.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | 1 mg Baricitinib | 2 mg Baricitinib
Number analyzed (Participants) | 146 | 147 | 145
percentage of participants | 5.5 | 4.1 | 4.1
Statistical Analysis 1: Comparison: Placebo vs 1 mg Baricitinib; Test type: Superiority; p = 0.598, Fisher Exact
Statistical Analysis 2: Comparison: Placebo vs 2 mg Baricitinib; Test type: Superiority; p = 0.785, Fisher Exact

16. Secondary Outcome: Percent Change From Baseline in Itch NRS
Description: The Itch NRS is a participant-administered, 11-point horizontal scale, with 0 representing "no itch" and 10 representing "worst itch imaginable." Overall severity of a participant's itching is indicated by selecting the number, using a daily diary, that best describes the worst level of itching in the past 24 hours.
  LS Means were calculated using a MMRM model with treatment, baseline disease severity (IGA),and treatment-by-visit-interaction as fixed categorical effects and baseline, and baseline-by-visit-interaction as fixed continuous effects.
Time Frame: Baseline, Week 16
Population: All randomized participants with Week 16 Itch NRS data.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo | 1 mg Baricitinib | 2 mg Baricitinib
Number analyzed (Participants) | 36 | 64 | 73
percent change | -18.01 (5.133) | -30.28 (4.104) | -39.87 (3.904)
Statistical Analysis 1: Comparison: Placebo vs 1 mg Baricitinib; Test type: Superiority; p = 0.063, Mixed Models Analysis; Mean Difference (Final Values) = -12.27, 95% CI 2-sided [-25.21 to 0.66], Standard Error of Mean 6.562
Statistical Analysis 2: Comparison: Placebo vs 2 mg Baricitinib; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = -21.85, 95% CI 2-sided [-34.54 to -9.17], Standard Error of Mean 6.437

17. Secondary Outcome: Change From Baseline in the Total Score of the Patient Oriented Eczema Measure (POEM)
Description: The POEM is a 7-item self-assessment questionnaire that assesses disease symptoms (dryness, itching, flaking, cracking, sleep loss, bleeding and weeping) on a scale ranging from 0-4 (0 = no days, 1 = 1-2 days, 2 = 3-4 days, 3 = 5-6 days, 4 = everyday). The sum of the 7 items gives the total POEM score of 0 (absent disease) to 28 (severe disease). High scores are indicative of more severe disease and poor quality of life.
  LS Means were calculated using a MMRM model with treatment, baseline disease severity (IGA), visit, and treatment-by-visit-interaction as fixed categorical effects and baseline and baseline-by-visit-interaction as fixed continuous effects.
Time Frame: Baseline, Week 16
Population: All randomized participants with Week 16 POEM data.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | 1 mg Baricitinib | 2 mg Baricitinib
Number analyzed (Participants) | 28 | 47 | 63
units on a scale | -2.67 (1.216) | -4.57 (0.937) | -7.44 (0.848)
Statistical Analysis 1: Comparison: Placebo vs 1 mg Baricitinib; Test type: Superiority; p = 0.217, Mixed Models Analysis; Mean Difference (Final Values) = -1.90, 95% CI 2-sided [-4.93 to 1.12], Standard Error of Mean 1.536
Statistical Analysis 2: Comparison: Placebo vs 2 mg Baricitinib; Test type: Superiority; p = 0.002, Mixed Models Analysis; Mean Difference (Final Values) = -4.77, 95% CI 2-sided [-7.70 to -1.84], Standard Error of Mean 1.487

18. Secondary Outcome: Change From Baseline in the Patient Global Impression of Severity-Atopic Dermatitis (PGI-S-AD) Score
Description: The PGI-S-AD is a single-item question asking the participant how they would rate their overall AD symptoms over the past 24 hours, using a daily diary. The 5 categories of responses are "(0) no symptoms", "(1) very mild", "(2) mild" "(3) moderate", and "(4) severe."
  LS Means were calculated using a MMRM model with treatment, baseline disease severity (IGA), visit, and treatment-by-visit-interaction as fixed categorical effects and baseline and baseline-by-visit-interaction as fixed continuous effects.
Time Frame: Baseline, Week 16
Population: All randomized participants with Week 16 PGI-S-AD data.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | 1 mg Baricitinib | 2 mg Baricitinib
Number analyzed (Participants) | 37 | 64 | 73
units on a scale | -0.46 (0.139) | -0.71 (0.111) | -0.88 (0.105)
Statistical Analysis 1: Comparison: Placebo vs 1 mg Baricitinib; Test type: Superiority; p = 0.155, Mixed Models Analysis; Mean Difference (Final Values) = -0.25, 95% CI 2-sided [-0.60 to 0.10], Standard Error of Mean 0.178
Statistical Analysis 2: Comparison: Placebo vs 2 mg Baricitinib; Test type: Superiority; p = 0.017, Mixed Models Analysis; Mean Difference (Final Values) = -0.42, 95% CI 2-sided [-0.76 to -0.07], Standard Error of Mean 0.174

19. Secondary Outcome: Change From Baseline on the Hospital Anxiety Depression Scale (HADS)
Description: The HADS is a participant-rated instrument used to assess both anxiety and depression. This instrument consists of 14 item questionnaire, each item is rated on a 4-point scale, giving maximum scores of 21 for anxiety and depression. Scores of 11 or more on either subscale are considered to be a significant 'case' of psychological morbidity, while scores of 8-10 represent 'borderline' and 0-7, 'normal.'
  LS Means were calculated using a MMRM model with treatment, baseline disease severity (IGA), visit, and treatment-by-visit-interaction as fixed categorical effects and baseline and baseline-by-visit-interaction as fixed continuous effects.
Time Frame: Baseline, Week 16
Population: All randomized participants with Week 16 HADS data.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | 1 mg Baricitinib | 2 mg Baricitinib
Number analyzed (Participants) | 28 | 47 | 63
units on a scale
  Anxiety | -2.03 (0.441) | -1.50 (0.356) | -2.55 (0.321)
  Depression | -1.31 (0.362) | -0.87 (0.294) | -1.73 (0.263)
Statistical Analysis 1: Comparison: Placebo vs 1 mg Baricitinib; Anxiety; Test type: Superiority; p = 0.345, Mixed Models Analysis; Mean Difference (Final Values) = 0.53, 95% CI 2-sided [-0.58 to 1.65], Standard Error of Mean 0.565
Statistical Analysis 2: Comparison: Placebo vs 2 mg Baricitinib; Anxiety; Test type: Superiority; p = 0.336, Mixed Models Analysis; Mean Difference (Final Values) = -0.52, 95% CI 2-sided [-1.59 to 0.55], Standard Error of Mean 0.543
Statistical Analysis 3: Comparison: Placebo vs 1 mg Baricitinib; Depression; Test type: Superiority; p = 0.353, Mixed Models Analysis; Mean Difference (Final Values) = 0.43, 95% CI 2-sided [-0.48 to 1.35], Standard Error of Mean 0.465
Statistical Analysis 4: Comparison: Placebo vs 2 mg Baricitinib; Depression; Test type: Superiority; p = 0.340, Mixed Models Analysis; Mean Difference (Final Values) = -0.43, 95% CI 2-sided [-1.31 to 0.45], Standard Error of Mean 0.446

20. Secondary Outcome: Change From Baseline on the Dermatology Life Quality Index (DLQI)
Description: The DLQI is a simple, participant-administered,10 question, validated, quality-of-life questionnaire that covers 6 domains including symptoms and feelings, daily activities, leisure, work and school, personal relationships, and treatment. The recall period of this scale is over the last "week." Response categories include "not at all," "a little," "a lot," and "very much," with corresponding scores of 0, 1, 2, and 3, respectively, and unanswered or "not relevant" responses scored as "0." Scores range from 0 to 30 ("no impact on participant's life" to "extremely large effect on participant's life"), and a 4-point change from baseline is considered as the minimal clinically important difference threshold.
  LS Means were calculated using a MMRM model with treatment, baseline disease severity (IGA),visit, and treatment-by-visit-interaction as fixed categorical and baseline, and baseline-by-visit-interaction as fixed continuous effects.
Time Frame: Baseline, Week 16
Population: All randomized participants with Week 16 DLQI data.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | 1 mg Baricitinib | 2 mg Baricitinib
Number analyzed (Participants) | 28 | 47 | 63
units on a scale | -3.97 (0.959) | -5.47 (0.776) | -7.46 (0.695)
Statistical Analysis 1: Comparison: Placebo vs 1 mg Baricitinib; Test type: Superiority; p = 0.224, Mixed Models Analysis; Mean Difference (Final Values) = -1.50, 95% CI 2-sided [-3.92 to 0.92], Standard Error of Mean 1.228
Statistical Analysis 2: Comparison: Placebo vs 2 mg Baricitinib; Test type: Superiority; p = 0.004, Mixed Models Analysis; Mean Difference (Final Values) = -3.50, 95% CI 2-sided [-5.83 to -1.16], Standard Error of Mean 1.184

21. Secondary Outcome: Change From Baseline on the Work Productivity and Activity Impairment - Atopic Dermatitis (WPAI-AD) Questionnaire
Description: The WPAI-AD participant questionnaire was developed to measure the effect of general health and symptom severity on work productivity and regular activities in the 7 days prior to the visit. The WPAI-AD consists of 6 items grouped in 4 domains: absenteeism (work time missed), presenteeism (impairment at work/reduced on-the-job effectiveness), work productivity loss (overall work impairment/absenteeism plus presenteeism), and activity impairment, that range from 0% to 100%, with higher values indicating greater impairment.
  LS Mean were calculated using a MMRM model with treatment, baseline disease severity (IGA), visit, and treatment-by-visit-interaction as fixed categorical effects and baseline and baseline-by-visit-interaction as fixed continuous effects.
Time Frame: Baseline, Week 16
Population: All randomized participants with baseline and at least 1 post-baseline WPAI measure.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | 1 mg Baricitinib | 2 mg Baricitinib
Number analyzed (Participants) | 28 | 47 | 62
units on a scale
  Absenteeism: number analyzed (Participants) | 16 | 27 | 41
  Absenteeism | 3.41 (4.741) | 0.05 (3.642) | 2.34 (3.078)
  Presenteeism: number analyzed (Participants) | 16 | 27 | 39
  Presenteeism | -3.44 (4.037) | -15.18 (3.315) | -19.33 (2.990)
  Overall Work Impairment: number analyzed (Participants) | 16 | 27 | 39
  Overall Work Impairment | -0.88 (4.848) | -13.73 (3.943) | -17.15 (3.520)
  Activity Impairment | -9.24 (3.334) | -18.87 (2.631) | -22.53 (2.401)
Statistical Analysis 1: Comparison: Placebo vs 1 mg Baricitinib; Absenteeism Change from Baseline; Test type: Superiority; p = 0.575, Mixed Models Analysis; Mean Difference (Final Values) = -3.36, 95% CI 2-sided [-15.30 to 8.57], Standard Error of Mean 5.956
Statistical Analysis 2: Comparison: Placebo vs 2 mg Baricitinib; Absenteeism Change from Baseline; Test type: Superiority; p = 0.851, Mixed Models Analysis; Mean Difference (Final Values) = -1.07, 95% CI 2-sided [-12.43 to 10.30], Standard Error of Mean 5.664
Statistical Analysis 3: Comparison: Placebo vs 1 mg Baricitinib; Presenteeism Change from Baseline; Test type: Superiority; p = 0.026, Mixed Models Analysis; Mean Difference (Final Values) = -11.75, 95% CI 2-sided [-22.05 to -1.45], Standard Error of Mean 5.212
Statistical Analysis 4: Comparison: Placebo vs 2 mg Baricitinib; Presenteeism Change from Baseline; Test type: Superiority; p = 0.002, Mixed Models Analysis; Mean Difference (Final Values) = -15.90, 95% CI 2-sided [-25.89 to -5.91], Standard Error of Mean 5.056
Statistical Analysis 5: Comparison: Placebo vs 1 mg Baricitinib; Overall Work Impairment Change from Baseline; Test type: Superiority; p = 0.041, Mixed Models Analysis; Mean Difference (Final Values) = -12.85, 95% CI 2-sided [-25.18 to -0.51], Standard Error of Mean 6.237
Statistical Analysis 6: Comparison: Placebo vs 2 mg Baricitinib; Overall Work Impairment Change from Baseline; Test type: Superiority; p = 0.008, Mixed Models Analysis; Mean Difference (Final Values) = -16.27, 95% CI 2-sided [-28.20 to -4.34], Standard Error of Mean 6.034
Statistical Analysis 7: Comparison: Placebo vs 1 mg Baricitinib; Activity Impairment Change from Baseline; Test type: Superiority; p = 0.023, Mixed Models Analysis; Mean Difference (Final Values) = -9.64, 95% CI 2-sided [-17.95 to -1.32], Standard Error of Mean 4.219
Statistical Analysis 8: Comparison: Placebo vs 2 mg Baricitinib; Activity Impairment Change from Baseline; Test type: Superiority; p = 0.001, Mixed Models Analysis; Mean Difference (Final Values) = -13.29, 95% CI 2-sided [-21.40 to -5.17], Standard Error of Mean 4.115

22. Secondary Outcome: Change From Baseline on the European Quality of Life-5 Dimensions 5 Levels (EQ-5D-5L) Index Score United States (US) and United Kingdom (UK) Algorithm
Description: The EQ-5D-5L is a 2-part measurement. The first part is comprised of the following 5 participant-reported dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems, and extreme problems. The responses are used to derive the health state index scores using the UK algorithm, with scores ranging from -0.594 to 1, and the US algorithm, with scores ranging from -0.109 to 1, with higher score indicating better health state.
  LS Means were calculated using a MMRM model with treatment, baseline disease activity (IGA), visit, and treatment-by-visit-interaction as fixed categorical effects and baseline and baseline-by-visit-interactions as fixed continuous effects.
Time Frame: Baseline, Week 16
Population: All randomized participants with Week 16 EQ-5D-5L Index Score US and UK Algorithm
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | 1 mg Baricitinib | 2 mg Baricitinib
Number analyzed (Participants) | 28 | 47 | 62
units on a scale
  Health State Index (US Algorithm) | 0.04 (0.021) | 0.06 (0.016) | 0.10 (0.015)
  Health State Index (UK Algorithm) | 0.07 (0.029) | 0.09 (0.023) | 0.14 (0.020)
Statistical Analysis 1: Comparison: Placebo vs 1 mg Baricitinib; Health State Index Score (US algorithm); Test type: Superiority; p = 0.482, Mixed Models Analysis; Mean Difference (Final Values) = 0.02, 95% CI 2-sided [-0.03 to 0.07], Standard Error of Mean 0.026
Statistical Analysis 2: Comparison: Placebo vs 2 mg Baricitinib; Health State Index Score (US algorithm); Test type: Superiority; p = 0.043, Mixed Models Analysis; Mean Difference (Final Values) = 0.05, 95% CI 2-sided [0.00 to 0.10], Standard Error of Mean 0.026
Statistical Analysis 3: Comparison: Placebo vs 1 mg Baricitinib; Health State Index Score (UK algorithm); Test type: Superiority; p = 0.656, Mixed Models Analysis; Mean Difference (Final Values) = 0.02, 95% CI 2-sided [-0.06 to 0.09], Standard Error of Mean 0.037
Statistical Analysis 4: Comparison: Placebo vs 2 mg Baricitinib; Health State Index Score (UK algorithm); Test type: Superiority; p = 0.057, Mixed Models Analysis; Mean Difference (Final Values) = 0.07, 95% CI 2-sided [-0.00 to 0.14], Standard Error of Mean 0.036

23. Secondary Outcome: Change From Baseline on the European Quality of Life-5 Dimensions 5 Levels (EQ-5D-5L) Visual Analog Score (VAS)
Description: EQ-5D-5L is a 2-part measurement. The second part is assessed using a visual analog scale (VAS) that ranges from 0 to 100 millimeter (mm), where 0 is the worst health you can imagine and 100 is the best health you can imagine.
  LS Means were calculated using a MMRM model with treatment, baseline disease activity (IGA), visit, and treatment-by-visit-interaction as fixed categorical effects and baseline and baseline-by-visit-interactions as fixed continuous effects.
Time Frame: Baseline, Week 16
Population: All randomized participants with Week 16 EQ-5D-5L VAS data.
Measure: Least Squares Mean (Standard Error); unit: millimeters
Arm/Group | Placebo | 1 mg Baricitinib | 2 mg Baricitinib
Number analyzed (Participants) | 28 | 47 | 62
millimeters | 4.67 (2.022) | 3.34 (1.631) | 8.14 (1.497)
Statistical Analysis 1: Comparison: Placebo vs 1 mg Baricitinib; Test type: Superiority; p = 0.609, Mixed Models Analysis; Mean Difference (Final Values) = -1.33, 95% CI 2-sided [-6.45 to 3.79], Standard Error of Mean 2.597
Statistical Analysis 2: Comparison: Placebo vs 2 mg Baricitinib; Test type: Superiority; p = 0.166, Mixed Models Analysis; Mean Difference (Final Values) = 3.48, 95% CI 2-sided [-1.46 to 8.41], Standard Error of Mean 2.503

24. Secondary Outcome: Percentage of Participants Achieving Investigator's Global Assessment (IGA) of 0 or 1 With a ≥ 2 Point Improvement
Description: as for outcome 2
Time Frame: Week 4
Population: All randomized participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | 1 mg Baricitinib | 2 mg Baricitinib
Number analyzed (Participants) | 147 | 147 | 146
percentage of participants | 2.7 [1.1 to 6.8] | 5.4 [2.8 to 10.4] | 8.2 [4.8 to 12.8]
Statistical Analysis 1: Comparison: Placebo vs 1 mg Baricitinib; Test type: Superiority; p = 0.258, Regression, Logistic; Odds Ratio (OR) = 1.96, 95% CI 2-sided [0.61 to 6.26]
Statistical Analysis 2: Comparison: Placebo vs 2 mg Baricitinib; Test type: Superiority; p = 0.052, Regression, Logistic; Odds Ratio (OR) = 2.99, 95% CI 2-sided [0.99 to 8.97]

ADVERSE EVENTS:
Time Frame: Baseline up to Week 104
Description: All randomized participants who receive at least 1 dose of investigational product and who did not discontinue from the study for the reason 'Lost to Follow-up' at the first post-baseline visit.
  Gender specific events only occurring in male or female participants have had the number of participants At Risk adjusted accordingly
Groups:
- Placebo (Period 1 WK 0 to 16): Placebo administered orally every day (Period 1 WK 0 to 16)
- 1 Milligram (mg) Baricitinib (Period 1 WK 0 to 16): 1 mg Baricitinib administered orally every day. Placebo administered orally to maintain the blind. (Period 1 WK 0 to 16)
- 2 mg Baricitinib (Period 1 WK 0 to 16): 2 mg Baricitinib administered orally every day. Placebo administered orally to maintain the blind. (Period 1 WK 0 to 16)
- Placebo (Period 2 WK 16 to 104): Placebo administered orally every day (Period 2 WK 16 to 104)
- 1 mg Baricitinib (Period 2 WK 16 to 104): 1 mg Baricitinib administered orally every day. Placebo administered orally to maintain the blind. (Period 2 WK 16 to 104)
- 2 mg Baricitinib (Period 2 WK 16 to 104): 2 mg Baricitinib administered orally every day. Placebo administered orally to maintain the blind. (Period 2 WK 16 to 104)
Arm/Group | Placebo (Period 1 WK 0 to 16) | 1 Milligram (mg) Baricitinib (Period 1 WK 0 to 16) | 2 mg Baricitinib (Period 1 WK 0 to 16) | Placebo (Period 2 WK 16 to 104) | 1 mg Baricitinib (Period 2 WK 16 to 104) | 2 mg Baricitinib (Period 2 WK 16 to 104)
All-Cause Mortality (participants affected / at risk) | 0/146 | 0/147 | 0/145 | 0/8 | 0/19 | 0/35
Serious Adverse Events (participants affected / at risk) | 3/146 | 1/147 | 2/145 | 0/8 | 0/19 | 0/35
Other Adverse Events (participants affected / at risk) | 34/146 | 24/147 | 36/145 | 1/8 | 10/19 | 11/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (Period 1 WK 0 to 16) (N=146) | 1 Milligram (mg) Baricitinib (Period 1 WK 0 to 16) (N=147) | 2 mg Baricitinib (Period 1 WK 0 to 16) (N=145) | Placebo (Period 2 WK 16 to 104) (N=8) | 1 mg Baricitinib (Period 2 WK 16 to 104) (N=19) | 2 mg Baricitinib (Period 2 WK 16 to 104) (N=35)
Hypertrophic cardiomyopathy (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Delusion (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hallucination (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Placebo (Period 1 WK 0 to 16) (N=146) | 1 Milligram (mg) Baricitinib (Period 1 WK 0 to 16) (N=147) | 2 mg Baricitinib (Period 1 WK 0 to 16) (N=145) | Placebo (Period 2 WK 16 to 104) (N=8) | 1 mg Baricitinib (Period 2 WK 16 to 104) (N=19) | 2 mg Baricitinib (Period 2 WK 16 to 104) (N=35)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 3 (3) | 6 (7) | 0 (0) | 0 (0) | 2 (2)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Seasonal allergy (Immune system disorders) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Eczema herpeticum (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Impetigo (Infections and infestations) | 3 (3) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Kidney infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 11 (12) | 3 (3) | 9 (9) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Tooth infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 9 (11) | 9 (9) | 10 (11) | 0 (0) | 2 (2) | 3 (4)
Urinary tract infection (Infections and infestations) | 3 (3) | 1 (1) | 5 (5) | 0 (0) | 0 (0) | 3 (3)
Viral upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 1 (1) | 3 (3) | 2 (3) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/79 (0) | 0/75 (0) | 0/68 (0) | 0/2 (0) | 0/4 (0) | 1/11 (1)
Micturition urgency (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Ovarian cyst ruptured (Reproductive system and breast disorders) | 0/67 (0) | 0/72 (0) | 0/77 (0) | 0/6 (0) | 1/15 (1) | 0/24 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) | 2 (2) | 0 (0) | 1 (1) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Actinic keratosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sinus operation (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2019-10-10): https://cdn.clinicaltrials.gov/large-docs/81/NCT03435081/Prot_000.pdf
  • Statistical Analysis Plan (2021-08-30): https://cdn.clinicaltrials.gov/large-docs/81/NCT03435081/SAP_002.pdf